CLINICAL TRIAL: NCT03414086
Title: Predictor of Clinical Response to Acthar in Myositis: Phase II of Acthar Clinical Trial
Brief Title: Predictor of Clinical Response to Acthar in Myositis
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rohit Aggarwal, MD, Associate Professor, University of Pittsburgh
Other Study IDs: PRO16100125
Record Dates: First submitted 2018-01-22; First posted 2018-01-29 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Myositis; Dermatomyositis; Polymyositis
Keywords: PM; DM
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — We will be collecting serum, cells, and pax gene samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Myositis in Remission: Subjects who are in remission with their myositis diagnosis.
  Interventions: Other: Myositis in Remission
- Healthy Controls: Subjects who do not have a myositis diagnosis.
  Interventions: Other: Healthy Control

INTERVENTIONS:
Other: Healthy Control — Ten healthy adult patients evaluating serum, PBMC's, and RNA.
  Groups: Healthy Controls
Other: Myositis in Remission — Ten patients (four who have polymyositis, six dermatomyositis) from our database who are followed in the Myositis Center. We will collect serum, PBMC's, and RNA samples will be obtained at baseline and at six months. Remission is defined as a global myositis disease activity score less than or equal to 1 on the MDAAT assessments with no new immunosuppressive drug or glucocorticoid use and no increase in dose of either in the preceding year.
  Groups: Myositis in Remission

SUMMARY:
Comparing the clinical effects of Acthar Gel before and after treatment and compare it to patients with inactive disease.

DETAILED DESCRIPTION:
To compare the clinical impact of Acthar Gel at the cellular and molecular level before and after treatment and compare it to patients with inactive disease. The cohort of active myositis subjects are not actually enrolled in this study, but rather the data for those with active myositis will be obtained from a previously completed trial entitled "Efficacy and safety of Adenocorticotropic Hormone Gel in Refractory dermatomyositis and polymyositis".

ELIGIBILITY:
Inclusion Criteria:

* Healthy Controls:

  * An individual will be eligible to be a control subject if his/her age is 18 years or greater.
* Myositis Remission Control Group

  * Definite or probable PM or DM by Bohan and Peter criteria.
  * PM patients must either possess a myositis-associated autoantibody or undergo adjudication for confirmation of the PM diagnosis by consensus of two experts (Aggarwal or Oddis) to ensure non-PM patients are not enrolled. This step is necessary since there are well known mimics of PM.
  * Age is greater than or equal to 18 years
  * Remission of myositis as defined by a myositis disease global activity score <1 on the MDAAT and no new immunosuppressive or glucocorticoid therapy or dose change within one year.

Exclusion Criteria:

* Healthy Controls:

  * An existing diagnosis of a CTD
  * A potential immune compromised state, for example, treatment with immunosuppressant or anti-rejection medication or a diagnosis of an immune deficiency disease
* Myositis Remission Control Group:

  * Juvenile DM or PM, myositis in overlap with another connective tissue disease, cancer associated myositis, inclusion body myositis, or any other non immune mediated myopathy.
  * Severe muscle damage defined as a baseline global muscle damage score on the MDI (Myositis Damage Index) of greater than or equal to five centimeters on a ten centimeter VAS.
  * Patients with malignancy within three years of screening (except basal cell cancer or squamous cell cancer of skin.
  * Uncontrolled diabetes, hepatic or renal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Arthritis and Autoimmunity Center
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2022-07-30 (Actual)

PRIMARY OUTCOMES:
IMACS Core Set Measures Improvement | 6 Months
  The International Myositis Assessment & Clinical Studies (IMACS) definition of improvement: Three of any of the six core set measures improved by greater than or equal to twenty percent, with no more than two core set measuring by greater than or equal to twenty five percent.

SECONDARY OUTCOMES:
Myositis Response Criteria | 6 Months
  This criteria yields a continuous improvement score which can be more readily extrapolated to individual response in subjects allowing correlation with baseline and longitudinal immunologic markers in these subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Aggarwal, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Outside researchers could obtain de-identified raw research data once approved from an ancillary committee.
Supporting Information: Study Protocol
Time Frame: Data will not be made available until afte the primary manuscript is published. Data will be available indefinitely.
Access Criteria: Approval from an ancillary committee.

REFERENCES:
- [Background] Bernstein RM, Morgan SH, Chapman J, Bunn CC, Mathews MB, Turner-Warwick M, Hughes GR. Anti-Jo-1 antibody: a marker for myositis with interstitial lung disease. Br Med J (Clin Res Ed). 1984 Jul 21;289(6438):151-2. doi: 10.1136/bmj.289.6438.151. PMID 6430389
- [Background] Catania A, Gatti S, Colombo G, Lipton JM. Targeting melanocortin receptors as a novel strategy to control inflammation. Pharmacol Rev. 2004 Mar;56(1):1-29. doi: 10.1124/pr.56.1.1. PMID 15001661
- [Background] Catania A, Lonati C, Sordi A, Carlin A, Leonardi P, Gatti S. The melanocortin system in control of inflammation. ScientificWorldJournal. 2010 Sep 14;10:1840-53. doi: 10.1100/tsw.2010.173. PMID 20852827
- [Background] Baram TZ, Mitchell WG, Tournay A, Snead OC, Hanson RA, Horton EJ. High-dose corticotropin (ACTH) versus prednisone for infantile spasms: a prospective, randomized, blinded study. Pediatrics. 1996 Mar;97(3):375-9. PMID 8604274
- [Background] Bomback AS, Tumlin JA, Baranski J, Bourdeau JE, Besarab A, Appel AS, Radhakrishnan J, Appel GB. Treatment of nephrotic syndrome with adrenocorticotropic hormone (ACTH) gel. Drug Des Devel Ther. 2011 Mar 14;5:147-53. doi: 10.2147/DDDT.S17521. PMID 21448451
- [Background] Simsarian JP, Saunders C, Smith DM. Five-day regimen of intramuscular or subcutaneous self-administered adrenocorticotropic hormone gel for acute exacerbations of multiple sclerosis: a prospective, randomized, open-label pilot trial. Drug Des Devel Ther. 2011;5:381-9. doi: 10.2147/DDDT.S19331. Epub 2011 Jul 11. PMID 21792296
- [Background] Levine T. Treating refractory dermatomyositis or polymyositis with adrenocorticotropic hormone gel: a retrospective case series. Drug Des Devel Ther. 2012;6:133-9. doi: 10.2147/DDDT.S33110. Epub 2012 Jun 11. PMID 22787386
- [Background] Page G, Chevrel G, Miossec P. Anatomic localization of immature and mature dendritic cell subsets in dermatomyositis and polymyositis: Interaction with chemokines and Th1 cytokine-producing cells. Arthritis Rheum. 2004 Jan;50(1):199-208. doi: 10.1002/art.11428. PMID 14730617
- [Background] Tournadre A, Lenief V, Eljaafari A, Miossec P. Immature muscle precursors are a source of interferon-beta in myositis: role of Toll-like receptor 3 activation and contribution to HLA class I up-regulation. Arthritis Rheum. 2012 Feb;64(2):533-41. doi: 10.1002/art.33350. PMID 22094963
- [Background] Tournadre A, Porcherot M, Cherin P, Marie I, Hachulla E, Miossec P. Th1 and Th17 balance in inflammatory myopathies: interaction with dendritic cells and possible link with response to high-dose immunoglobulins. Cytokine. 2009 Jun;46(3):297-301. doi: 10.1016/j.cyto.2009.02.013. Epub 2009 Mar 19. PMID 19303320
- [Background] Acosta-Rodriguez EV, Napolitani G, Lanzavecchia A, Sallusto F. Interleukins 1beta and 6 but not transforming growth factor-beta are essential for the differentiation of interleukin 17-producing human T helper cells. Nat Immunol. 2007 Sep;8(9):942-9. doi: 10.1038/ni1496. Epub 2007 Aug 5. PMID 17676045
- [Background] McGeachy MJ, Cua DJ. The link between IL-23 and Th17 cell-mediated immune pathologies. Semin Immunol. 2007 Dec;19(6):372-6. doi: 10.1016/j.smim.2007.10.012. Epub 2007 Dec 3. PMID 18319054
- [Background] Chevrel G, Page G, Granet C, Streichenberger N, Varennes A, Miossec P. Interleukin-17 increases the effects of IL-1 beta on muscle cells: arguments for the role of T cells in the pathogenesis of myositis. J Neuroimmunol. 2003 Apr;137(1-2):125-33. doi: 10.1016/s0165-5728(03)00032-8. PMID 12667656
- [Background] Tournadre A, Lenief V, Miossec P. Expression of Toll-like receptor 3 and Toll-like receptor 7 in muscle is characteristic of inflammatory myopathy and is differentially regulated by Th1 and Th17 cytokines. Arthritis Rheum. 2010 Jul;62(7):2144-51. doi: 10.1002/art.27465. PMID 20309865
- [Background] Bilgic H, Ytterberg SR, Amin S, McNallan KT, Wilson JC, Koeuth T, Ellingson S, Newman B, Bauer JW, Peterson EJ, Baechler EC, Reed AM. Interleukin-6 and type I interferon-regulated genes and chemokines mark disease activity in dermatomyositis. Arthritis Rheum. 2009 Nov;60(11):3436-46. doi: 10.1002/art.24936. PMID 19877033
- [Background] Scuderi F, Mannella F, Marino M, Provenzano C, Bartoccioni E. IL-6-deficient mice show impaired inflammatory response in a model of myosin-induced experimental myositis. J Neuroimmunol. 2006 Jul;176(1-2):9-15. doi: 10.1016/j.jneuroim.2006.03.026. Epub 2006 May 24. PMID 16725212
- [Background] Okiyama N, Sugihara T, Iwakura Y, Yokozeki H, Miyasaka N, Kohsaka H. Therapeutic effects of interleukin-6 blockade in a murine model of polymyositis that does not require interleukin-17A. Arthritis Rheum. 2009 Aug;60(8):2505-12. doi: 10.1002/art.24689. PMID 19644888
- [Background] Narazaki M, Hagihara K, Shima Y, Ogata A, Kishimoto T, Tanaka T. Therapeutic effect of tocilizumab on two patients with polymyositis. Rheumatology (Oxford). 2011 Jul;50(7):1344-6. doi: 10.1093/rheumatology/ker152. Epub 2011 Apr 22. No abstract available. PMID 21515628
- [Background] Grogan JL, Ouyang W. A role for Th17 cells in the regulation of tertiary lymphoid follicles. Eur J Immunol. 2012 Sep;42(9):2255-62. doi: 10.1002/eji.201242656. PMID 22949324
- [Background] Patakas A, Benson RA, Withers DR, Conigliaro P, McInnes IB, Brewer JM, Garside P. Th17 effector cells support B cell responses outside of germinal centres. PLoS One. 2012;7(11):e49715. doi: 10.1371/journal.pone.0049715. Epub 2012 Nov 16. PMID 23166752
- [Background] Ma CS, Deenick EK, Batten M, Tangye SG. The origins, function, and regulation of T follicular helper cells. J Exp Med. 2012 Jul 2;209(7):1241-53. doi: 10.1084/jem.20120994. PMID 22753927
- [Background] Ma CS, Deenick EK. Human T follicular helper (Tfh) cells and disease. Immunol Cell Biol. 2014 Jan;92(1):64-71. doi: 10.1038/icb.2013.55. Epub 2013 Oct 22. PMID 24145858
- [Background] Diehl SA, Schmidlin H, Nagasawa M, Blom B, Spits H. IL-6 triggers IL-21 production by human CD4+ T cells to drive STAT3-dependent plasma cell differentiation in B cells. Immunol Cell Biol. 2012 Sep;90(8):802-11. doi: 10.1038/icb.2012.17. Epub 2012 Apr 10. PMID 22491065
- [Background] Dienz O, Eaton SM, Bond JP, Neveu W, Moquin D, Noubade R, Briso EM, Charland C, Leonard WJ, Ciliberto G, Teuscher C, Haynes L, Rincon M. The induction of antibody production by IL-6 is indirectly mediated by IL-21 produced by CD4+ T cells. J Exp Med. 2009 Jan 16;206(1):69-78. doi: 10.1084/jem.20081571. Epub 2009 Jan 12. PMID 19139170
- [Background] Kimura A, Kishimoto T. IL-6: regulator of Treg/Th17 balance. Eur J Immunol. 2010 Jul;40(7):1830-5. doi: 10.1002/eji.201040391. PMID 20583029
- [Background] Carbone G, Wilson A, Diehl SA, Bunn J, Cooper SM, Rincon M. Interleukin-6 receptor blockade selectively reduces IL-21 production by CD4 T cells and IgG4 autoantibodies in rheumatoid arthritis. Int J Biol Sci. 2013;9(3):279-88. doi: 10.7150/ijbs.5996. Epub 2013 Mar 7. PMID 23493630
- [Background] Morita R, Schmitt N, Bentebibel SE, Ranganathan R, Bourdery L, Zurawski G, Foucat E, Dullaers M, Oh S, Sabzghabaei N, Lavecchio EM, Punaro M, Pascual V, Banchereau J, Ueno H. Human blood CXCR5(+)CD4(+) T cells are counterparts of T follicular cells and contain specific subsets that differentially support antibody secretion. Immunity. 2011 Jan 28;34(1):108-21. doi: 10.1016/j.immuni.2010.12.012. Epub 2011 Jan 6. PMID 21215658
- [Background] Baechler EC, Bilgic H, Reed AM. Type I interferon pathway in adult and juvenile dermatomyositis. Arthritis Res Ther. 2011;13(6):249. doi: 10.1186/ar3531. Epub 2011 Dec 22. PMID 22192711
- [Background] Sweeney CM, Lonergan R, Basdeo SA, Kinsella K, Dungan LS, Higgins SC, Kelly PJ, Costelloe L, Tubridy N, Mills KH, Fletcher JM. IL-27 mediates the response to IFN-beta therapy in multiple sclerosis patients by inhibiting Th17 cells. Brain Behav Immun. 2011 Aug;25(6):1170-81. doi: 10.1016/j.bbi.2011.03.007. Epub 2011 Mar 21. PMID 21420486
- [Background] Biswas PS, Aggarwal R, Levesque MC, Maers K, Ramani K. Type I interferon and T helper 17 cells co-exist and co-regulate disease pathogenesis in lupus patients. Int J Rheum Dis. 2015 Jul;18(6):646-53. doi: 10.1111/1756-185X.12636. Epub 2015 May 11. PMID 25960196
- [Background] Gunawardena H, Betteridge ZE, McHugh NJ. Myositis-specific autoantibodies: their clinical and pathogenic significance in disease expression. Rheumatology (Oxford). 2009 Jun;48(6):607-12. doi: 10.1093/rheumatology/kep078. PMID 19439503
- [Background] Aggarwal R, Cassidy E, Fertig N, Koontz DC, Lucas M, Ascherman DP, Oddis CV. Patients with non-Jo-1 anti-tRNA-synthetase autoantibodies have worse survival than Jo-1 positive patients. Ann Rheum Dis. 2014 Jan;73(1):227-32. doi: 10.1136/annrheumdis-2012-201800. Epub 2013 Feb 19. PMID 23422076
- [Background] rohit aggarwal cvo, andriy bandos, Danielle goudeau, diane koontz, qi zenbiao, ann m. reed. dan p ascherman, and marc c levesque. . effect of b cell depletion therapy with rituximab on myositis associated antibody levels in idiopathic inflammatory myopathy. arthritis and research. 2012;64(10(suppl.)):s325.
- [Background] Greenberg SA, Bradshaw EM, Pinkus JL, Pinkus GS, Burleson T, Due B, Bregoli L, O'Connor KC, Amato AA. Plasma cells in muscle in inclusion body myositis and polymyositis. Neurology. 2005 Dec 13;65(11):1782-7. doi: 10.1212/01.wnl.0000187124.92826.20. PMID 16344523
- [Background] Khanna S, Reed AM. Immunopathogenesis of juvenile dermatomyositis. Muscle Nerve. 2010 May;41(5):581-92. doi: 10.1002/mus.21669. PMID 20405498
- [Background] Karnowski A, Chevrier S, Belz GT, Mount A, Emslie D, D'Costa K, Tarlinton DM, Kallies A, Corcoran LM. B and T cells collaborate in antiviral responses via IL-6, IL-21, and transcriptional activator and coactivator, Oct2 and OBF-1. J Exp Med. 2012 Oct 22;209(11):2049-64. doi: 10.1084/jem.20111504. Epub 2012 Oct 8. PMID 23045607
- [Background] Kishimoto T. Interleukin-6: discovery of a pleiotropic cytokine. Arthritis Res Ther. 2006;8 Suppl 2(Suppl 2):S2. doi: 10.1186/ar1916. Epub 2006 Jul 28. PMID 16899106
- [Background] Sweet RA, Lee SK, Vinuesa CG. Developing connections amongst key cytokines and dysregulated germinal centers in autoimmunity. Curr Opin Immunol. 2012 Dec;24(6):658-64. doi: 10.1016/j.coi.2012.10.003. Epub 2012 Nov 1. PMID 23123277
- [Background] Oddis CV, Reed AM, Aggarwal R, Rider LG, Ascherman DP, Levesque MC, Barohn RJ, Feldman BM, Harris-Love MO, Koontz DC, Fertig N, Kelley SS, Pryber SL, Miller FW, Rockette HE; RIM Study Group. Rituximab in the treatment of refractory adult and juvenile dermatomyositis and adult polymyositis: a randomized, placebo-phase trial. Arthritis Rheum. 2013 Feb;65(2):314-24. doi: 10.1002/art.37754. PMID 23124935
- [Background] Aggarwal R, Bandos A, Reed AM, Ascherman DP, Barohn RJ, Feldman BM, Miller FW, Rider LG, Harris-Love MO, Levesque MC; RIM Study Group; Oddis CV. Predictors of clinical improvement in rituximab-treated refractory adult and juvenile dermatomyositis and adult polymyositis. Arthritis Rheumatol. 2014 Mar;66(3):740-9. doi: 10.1002/art.38270. PMID 24574235
- [Background] Aggarwal R, Oddis CV, Goudeau D, Fertig N, Metes I, Stephens C, Qi Z, Koontz D, Levesque MC. Anti-signal recognition particle autoantibody ELISA validation and clinical associations. Rheumatology (Oxford). 2015 Jul;54(7):1194-9. doi: 10.1093/rheumatology/keu436. Epub 2014 Dec 17. PMID 25524922
- [Background] aggarwal r oc, bandos a, goudeau d, koontz d, zenbia q, reed am, ascherman dp, levesque mc. effect of b cell depletion therapy with rituximab on myositis associated antibody levels in idiopathic inflammatory myopathy. arthritis and research. 2012;64(10(suppl)):s325.
- [Background] aggarwal r oc, Wilkerson er, koontz d, metes id, reed am, ascherman dp, levesque mc. peripheral blood memory b cell numbers predit clinical response following rituximab treatment of adult and childhood myositis. arthritis and research. 2013;65(10(suppl)):s755-66.
- [Background] Rider LG, Lachenbruch PA, Monroe JB, Ravelli A, Cabalar I, Feldman BM, Villalba ML, Myones BL, Pachman LM, Rennebohm RM, Reed AM, Miller FW; IMACS Group. Damage extent and predictors in adult and juvenile dermatomyositis and polymyositis as determined with the myositis damage index. Arthritis Rheum. 2009 Nov;60(11):3425-35. doi: 10.1002/art.24904. PMID 19877055
- [Background] Aggarwal R, Lucas M, Fertig N, Oddis CV, Medsger TA Jr. Anti-U3 RNP autoantibodies in systemic sclerosis. Arthritis Rheum. 2009 Apr;60(4):1112-8. doi: 10.1002/art.24409. PMID 19333934
- [Background] Rider LG, Werth VP, Huber AM, Alexanderson H, Rao AP, Ruperto N, Herbelin L, Barohn R, Isenberg D, Miller FW. Measures of adult and juvenile dermatomyositis, polymyositis, and inclusion body myositis: Physician and Patient/Parent Global Activity, Manual Muscle Testing (MMT), Health Assessment Questionnaire (HAQ)/Childhood Health Assessment Questionnaire (C-HAQ), Childhood Myositis Assessment Scale (CMAS), Myositis Disease Activity Assessment Tool (MDAAT), Disease Activity Score (DAS), Short Form 36 (SF-36), Child Health Questionnaire (CHQ), physician global damage, Myositis Damage Index (MDI), Quantitative Muscle Testing (QMT), Myositis Functional Index-2 (FI-2), Myositis Activities Profile (MAP), Inclusion Body Myositis Functional Rating Scale (IBMFRS), Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI), Cutaneous Assessment Tool (CAT), Dermatomyositis Skin Severity Index (DSSI), Skindex, and Dermatology Life Quality Index (DLQI). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S118-57. doi: 10.1002/acr.20532. No abstract available. PMID 22588740